CLINICAL TRIAL: NCT00783237
Title: Onset of Action of Mometasone Furoate Nasal Spray vs. Placebo in Induced Allergic Rhinitis
Brief Title: Onset of Effect of Mometasone Nasal Spray in Induced Allergic Rhinitis (Study P03431)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03431
Expanded Access: Available
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone Furoate Nasal Spray (Experimental)
  Interventions: Drug: Mometasone
- Placebo Nasal Spray (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone — Mometasone Furoate Nasal Spray, single dose of 200 mcg (2 sprays per nostril)
  Other Names: Nasonex, SCH 032088
  Arms: Mometasone Furoate Nasal Spray
Drug: Placebo — Placebo nasal spray, single dose of 2 sprays per nostril
  Arms: Placebo Nasal Spray

SUMMARY:
This was a single-dose study to determine the time it takes for mometasone furoate nasal spray to go in effect, after a single dose of 2 sprays per nostril. Patients who are eligible were exposed to ragweed pollen for 3 hours on one or two occasions. Patients who experienced adequate symptoms during the pollen exposure phase came back for a Treatment Phase visit. During the Treatment Phase visit, patients were exposed to ragweed pollen for 2 hours and then received either mometasone or placebo nasal spray. Symptom evaluations began on the patients every hour for the next 11 hours.

ELIGIBILITY:
Inclusion Criteria:

* at least 12 years old,
* had a history of SAR to ragweed pollen for at least one year
* had a positive skin test (prick) to short ragweed allergen.
* if female, had a negative urine pregnancy test (HCG) at the Screening Visit, and prior to treatment on the Treatment Visit
* were non pregnant women of childbearing potential and used a medically acceptable, adequate form of birth control.

Exclusion Criteria:

* developed signs or symptoms of bronchospasm, i.e., wheezing, dyspnea, and/or cough, during the priming sessions;
* had any significant medical condition which, in the judgment of the investigator, might interfere with the study or require treatment;
* had an upper respiratory or sinus infection within two weeks prior to treatment;
* had received escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy for treatment of rhinitis;
* were female subjects who were pregnant, breast feeding, or premenarchal;
* could not adhere to concomitant medication prohibitions;
* had a known potential for hypersensitivity, allergy, or idiosyncratic reaction to mometasone furoate nasal spray;
* had asthma that requires systemic or inhaled corticosteroid treatment;
* had large nasal polyps, marked septum deviations, or any other nasal structural abnormality that significantly interferes with nasal airflow;
* had rhinitis medicamentosa;
* had any relevant abnormal vital sign due to an unknown underlying disease and considered by the investigator and Sponsor Monitor to contraindicate study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2003-12-01 (Actual); Primary Completion 2004-02-21 (Actual); Study Completion 2004-02-21 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | On the day of treatment, after 90 and 120 minutes of pollen exposure and every 60 minutes post-dose for 12 hours

SECONDARY OUTCOMES:
Nasal and Non-Nasal symptoms, Total Nasal and Total Non-Nasal symptoms, Total Symptom Score, Global Therapeutic Response | On the day of treatment, after 90 and 120 minutes of pollen exposure and every 60 minutes post-dose for 12 hours

REFERENCES:
- [Result] Berger WE, Nayak AS, Staudinger HW. Mometasone furoate improves congestion in patients with moderate-to-severe seasonal allergic rhinitis. Ann Pharmacother. 2005 Dec;39(12):1984-9. doi: 10.1345/aph.1G202. Epub 2005 Nov 8. PMID 16278257